CLINICAL TRIAL: NCT01298531
Title: A Multi Centre, Double Blind, Placebo-controlled Study to Evaluate the Non Steroidal Anti-inflamatory Drugs (NSAIDS) Sparing Effect of Etanercept in Adult Subjects With Axial Involvement of Spondyloarthritis
Brief Title: A Study to Evaluate the NSAIDS Sparing Effect of Etanercept in Subjects With Axial Spondyloarthritis
Acronym: SPARSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1801132; 0881A1-4749
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Results first posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Axial Spondyloarthritis
Keywords: Etanercept; Axial Spondyloarthritis; NSAIDs sparing effect
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- etanercept (Active Comparator): Group A: etanercept 50 mg subcutaneous (SC) injections once weekly for 16 weeks.
  Interventions: Drug: etanercept
- etanercept-placebo (Placebo Comparator): Group B: placebo subcutaneous (SC) injections once weekly for (how many) weeks follwed by etanercept 50 mg SC injections once weekly.
  Interventions: Drug: etanercept; Drug: placebo

INTERVENTIONS:
Drug: etanercept — etanercept 50 mg subcutaneous (SC) injections once weekly for 16 weeks.
  Other Names: Enbrel
  Arms: etanercept
Drug: etanercept — etanercept 50 mg subcutaneous (SC) injections once weekly for 8 weeks following the prior 8 weeks of placebo.
  Other Names: Enbrel
  Arms: etanercept-placebo
Drug: placebo — placebo subcutaneous (SC) injections once weekly for 8 weeks.
  Arms: etanercept-placebo

SUMMARY:
This study will compare the Non Steroidal Anti-Inflammatory Drugs (NSAIDs) sparing effect of etanercept with that of placebo in adult subjects with axial Spondyloarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 years and over at the time of consent to the study.
* Diagnosis of SpA, as defined by the ASAS criteria for axial SpA
* Axial involvement refractory to previous or current intake of NSAIDs, defined as at least 2 NSAIDs at maximum tolerated dose determined from past medical history taken for a duration of > 1 month (for both NSAIDs combined) before the Screening visit.
* Active axial involvement defined by mini BASDAI

Exclusion Criteria:

* Subjects who are investigational site staff members or subjects who are Pfizer employees directly involved in the conduct of the trial.
* Subjects who have received any previous treatment with etanercept or other TNFα inhibitors or biologic agents.
* Subjects with a known or expected allergy, contraindication, or hypersensitivity to etanercept or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- France (19):
  - Institut Calot - Fondation Hopale, Berck, France
  - Hopital Pellegrin, Bordeaux
  - Centre Hospitalier, Service de Rhumatologie, Cahors
  - CHU Hopital Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - Chu Dupuytren, Rhumatologie et Therapeutique, Limoges
  - CHU Lapeyronie, Immuno-Rhumatologie, Montpellier
  - Hopital de l'Archet, Nice
  - Hopital Porte Madeleine, Orléans
  - H�al Saint-Antoine, Paris
  - Hopital Cochin, Paris
  - Hopital Saint Joseph - Service de Rhumatologie, Paris
  - Hopital Bichat, Paris
  - Service de Rhumatologie, Paris
  - CHU Bois Guillaume - Service de Rhumatologie, Rouen
  - CHU de Saint Etienne, Hopital Nord, Saint-Etienne
  - Hopital Purpan, Toulouse

REFERENCES:
- [Derived] Dougados M, Wood E, Gossec L, Dubanchet A, Logeart I, van der Heijde D. Discriminant Capacity of Clinical Efficacy and Nonsteroidal Antiinflammatory Drug-sparing Endpoints, Alone or in Combination, in Axial Spondyloarthritis. J Rheumatol. 2015 Dec;42(12):2361-8. doi: 10.3899/jrheum.150378. Epub 2015 Nov 15. PMID 26568588
- [Derived] Dougados M, Wood E, Combe B, Schaeverbeke T, Miceli-Richard C, Berenbaum F, Koppiker N, Dubanchet A, Logeart I. Evaluation of the nonsteroidal anti-inflammatory drug-sparing effect of etanercept in axial spondyloarthritis: results of the multicenter, randomized, double-blind, placebo-controlled SPARSE study. Arthritis Res Ther. 2014 Nov 27;16(6):481. doi: 10.1186/s13075-014-0481-5. PMID 25428762
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801132&StudyName=A%20Study%20to%20Evaluate%20the%20NSAIDS%20Sparing%20Effect%20of%20Etanercept%20in%20Subjects%20with%20Axial%20Spondyloarthritis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 128 screened participants, 90 were assigned to either double-blind etanercept (ETN) 50 mg to open-label ETN 50 mg or placebo to open-label ETN 50 mg group. Participants entered an escape arm at Week 4 visit if the total back pain or the BASDAI score increased >50% vs baseline or participants were with maximum tolerated NSAIDs.
Pre-assignment Details: Four participants who were randomized to receive placebo in the double-blind phase were withdrawn during this phase, and they did not enter the escape arm, so these four participants never received ETN.
Groups:
- Double Blind ETN 50 mg to Open Label ETN 50 mg Group: Participants were treated with ETN 50 mg subcutaneous injections once weekly for 16 weeks
- Placebo to Open Label ETN 50 mg Group: Participants were treated with Placebo subcutaneous injections once weekly for 8 weeks followed by ETN 50 mg SC injections once weekly for 8 weeks
Period: Overall Study
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Started | 42 | 48
Completed | 33 | 41
Not Completed | 9 | 7
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 4 | 3
Not completed — Does not meet entrance criteria | 0 | 1
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group | Total
Number analyzed (Participants) | 42 | 48 | 90
Age, Customized [Number; unit: Participants]
  18 - 44 Years | 31 | 32 | 63
  45 - 64 Years | 9 | 15 | 24
  ≥ 65 Years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 24 | 32 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Non Steroidal Anti Inflammatory Drug (NSAID) Assessment of the SpondyloArthritis International Society (ASAS) Score at Week 8.
Description: Diary data from the 7 days prior to respective visit were used to evaluate the endpoint, where the score was only calculated if at least 5 of the 7 days data were available. Score was calculated from NSAID usage completed on diary cards considering NSAID type, total daily dose and number of days consumed. The Daily diclofenac-equivalent dose score was derived by converting each daily dose of NSAID to a percentage dose equivalent of 150 mg diclofenac; e.g. 1000 mg naproxen is equivalent to 150 mg diclofenac. For each NSAID, the percentage diclofenac-equivalent score is then multiplied by daily dose frequency and proportion of the period where dose was taken.
  Ie Score=M x F x n/N (M: Percentage dose equivalent to diclofenac; F=Daily Dose Frequency; n=number of days with NSAID; N=number of days in period). The NSAID ASAS score is the sum of all such scores for all NSAIDs taken during the period. The minimum value is 0 and a higher NSAID-ASAS value indicates greater NSAIDs consumption.
Time Frame: Week 8
Population: The Intent To Treat (ITT) population comprised all participants who received at least one dose of the randomized treatment. Participants were analyzed according to treatment randomized and any data recorded after entry into the escape arm were included in the analysis. Missing data were imputed through last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 39 | 42
Scores on a scale | -63.90 (6.09) | -36.63 (5.87)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; The primary analysis of the primary endpoint was an Analysis of covariance (ANCOVA)with Baseline NSAID score and treatment as explanatory variables. The hypothesis tested for the primary endpoint was as follows: H0: ΔETN = ΔPlacebo; H1: ΔETN ≠ ΔPlacebo; Test type: Superiority or Other; p = 0.0019, ANCOVA; Not specifed; Mean Difference (Final Values) = -27.27, 95% CI 2-sided [-44.17 to -10.38]

2. Secondary Outcome: Total NSAID ASAS [Area Under Curve (AUC)] Score From Baseline to Week 8.
Description: The total NSAID score for the first 8 weeks of randomized treatment was calculated as an AUC using the linear trapezoidal rule. LOCF will only be applied where the subject is still in the study and the NSAID score is missing.
Time Frame: Week 8
Population: The ITT population comprised all participants who received at least one dose of the randomized treatment. Participants were analyzed according to treatment randomized and any data recorded after entry into the escape arm were included in the analysis. Missing data were imputed through LOCF approach.
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale * days
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 40 | 42
Unit on a scale * days | 45.24 (5.44) | 65.02 (5.30)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; The analysis of secondary endpoints was an ANCOVA using linear regression with Baseline NSAID score and MMRM was run using the model and using the repeated measures for the changes from Baseline in each outcome at Week 8; Test type: Superiority or Other; p = 0.0115, ANCOVA; Mean Difference (Final Values) = -19.78, 95% CI 2-sided [-34.99 to -4.57]

3. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 4.
Description: A numeric rating scale was used, for questions 1-5 (Fatigue, Spinal Pain, Joint pain or Swelling, Discomfort and Morning stiffness severity respectively) on a scale from 0 (none) to 10 (very severe). Question 6 (morning stiffness duration) was recorded on a scale of 0 (0 or more hours) to 10 (2 hours). To give the five major Ankylosing Spondylitis (AS) symptoms equal weighting, the average of the two scores relating to morning stiffness was taken. This averaged morning stiffness score was then summed with the remaining 4 questions, resulting in a composite score on a scale of 0-50, which was then divided by 5 to give the final BASDAI score on a scale of 0-10.
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 39 | 44
Units on a scale | -1.50 (0.27) | -0.56 (0.26)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; The analysis of secondary endpoints was an ANCOVA using linear regression with Baseline NSAID score and MMRM was run using the model as detailed for the primary endpoint and using the repeated measures for the changes from Baseline in each outcome at Week 4; Test type: Superiority or Other; p = 0.0153, ANCOVA; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-1.68 to -0.18]

4. Secondary Outcome: Change From Baseline in BASDAI at Week 8
Description: A numeric rating scale was used, for questions 1-5 (Fatigue, Spinal Pain, Joint pain or Swelling, Discomfort and Morning stiffness severity respectively) on a scale from 0 (none) to 10 (very severe). Question 6 (morning stiffness duration) was recorded on a scale of 0 (0 or more hours) to 10 (2 hours). To give the five major AS symptoms equal weighting, the average of the two scores relating to morning stiffness was taken. This averaged morning stiffness score was then summed with the remaining 4 questions, resulting in a composite score on a scale of 0-50, which was then divided by 5 to give the final BASDAI score on a scale of 0-10.
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 41 | 45
Units on a scale | -2.01 (0.32) | -1.13 (0.31)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; The analysis of secondary endpoints was an ANCOVA using linear regression with Baseline NSAID score and MMRM was run using the model as detailed for the primary endpoint and using the repeated measures for the changes from Baseline in each outcome at Week 8; Test type: Superiority or Other; p = 0.0510, ANCOVA; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-1.76 to 0.00]

5. Secondary Outcome: Change From Baseline in BASDAI Score at Weeks 12 and 16.
Description: as for outcome 4
Time Frame: Week 12 and 16
Population: The ITT population comprised all participants who received at least one dose of the randomized treatment. Participants were analyzed according to treatment randomized and any data recorded after entry into the escape arm were included in the analysis. This analysis was with the observed cases.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Units on a scale
  Week 12 (N=36, N=41) | -2.5 (2.35) | -2.6 (2.12)
  Week 16 (N=28, N=37) | -2.6 (1.83) | -3.0 (2.14)

6. Secondary Outcome: Number of Participants Using NSAIDs at Week 8.
Description: Participants who received NSAIDs at Week 8 were reported.
Time Frame: Week 8
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 33 | 40
Participants | 17 | 32
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; Logistic regression with baseline score and treatment group included as covariates; Test type: Superiority or Other; p = 0.0066, Regression, Logistic; Odds Ratio (OR) = 0.209, 95% CI 2-sided [0.07 to 0.65]

7. Secondary Outcome: Change From Baseline in Mini BASDAI at Week 8 (AUC).
Description: as for outcome 4
Time Frame: Week 8
Population: The ITT population comprised all participants who received at least one dose of the randomized treatment. The efficacy analysis was based on the ITT population. Participants were analyzed according to treatment randomized and any data recorded after entry into the escape arm were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale * days
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 41 | 46
Unit on a scale * days | 275.68 (13.64) | 329.37 (12.88)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; The changes from baseline in the continuous endpoints of mini BASDAI was analyzed using ANCOVA. The total NSAID score for the first 8 weeks of randomized treatment was calculated as an AUC using the linear trapezoidal rule; Test type: Superiority or Other; p = 0.0053, ANCOVA; Mean Difference (Final Values) = -53.70, 95% CI 2-sided [-91.01 to -16.38]

8. Secondary Outcome: Number of Participants Achieved BASDAI 50 at Week 8.
Description: Response was defined as a 50% improvement of the baseline BASDAI after 8 Weeks.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 41 | 45
Participants | 16 | 8
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; Logistic regression with baseline morning stiffness score and treatment group included as covariates; Test type: Superiority or Other; p = 0.0324, Regression, Logistic; Odds Ratio (OR) = 2.963, 95% CI 2-sided [1.10 to 8.01]

9. Secondary Outcome: Number of Participants Achieved BASDAI 50 at Weeks 4, 12 and 16.
Description: Response was defined as a 50% improvement of the baseline BASDAI after 4, 12 and 16 Weeks.
Time Frame: Weeks 4, 12 and 16
Population: The ITT population comprised all participants who received at least one dose of the randomized treatment. Participants were analyzed according to treatment randomized and any data recorded after entry into the escape arm were included in the analysis. This analysis was performed with the observed cases.
Measure: Number; unit: Participants
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Participants
  Week 4 (N=39, N=44) | 10 | 3
  Week 12 (N=36, N=41) | 17 | 19
  Week 16 (N=28, N=37) | 15 | 18

10. Secondary Outcome: Number of Participants Achieving ASAS 20 (Assessment of the Spondylo Arthritis International Society 20) at Weeks 4, 12 and 16
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) participants ASAS = 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 20 = 20% improvement from baseline and an absolute change ≥ 10 units on a 0-100 scale (0=no disease activity; 100=high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: Weeks 4, 12 and 16
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Participants
  Week 4 (N = 38, 42) | 14 | 5
  Week 12 (N = 35, 37) | 17 | 21
  Week 16 (N = 28, 36) | 18 | 23

11. Secondary Outcome: Number of Participants Achieving ASAS 20 at Week 8
Description: as for outcome 10
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 36 | 42
Participants | 16 | 10
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; Week 8 was analyzed using a logistic regression to assess treatment effect. Logistic regression with baseline morning stiffness score and treatment group included as covariates; Test type: Superiority or Other; p = 0.0501, Regression, Logistic; Odds Ratio (OR) = 2.696, 95% CI 2-sided [1.00 to 7.27]

12. Secondary Outcome: Number of Participants Achieving ASAS 40 at Weeks 4, 12 and 16.
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) participants ASAS = 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 40 = 40% improvement from baseline and an absolute change ≥ 20 units on a 0-100 scale (0=no disease activity, 100=high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: Weeks 4, 12 and 16
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Participants
  Week 4 (N = 38, 42) | 9 | 3
  Week 12 (N = 35, 37) | 17 | 20
  Week 16 (N = 28, 36) | 16 | 20

13. Secondary Outcome: Number of Participants Achieving ASAS 40 at Week 8
Description: as for outcome 12
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 36 | 42
Participants | 16 | 9
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.0284, Regression, Logistic; Odds Ratio (OR) = 3.103, 95% CI 2-sided [1.13 to 8.54]

14. Secondary Outcome: Number of Participants Achieving ASAS 70 at Weeks 4, 12 and 16.
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) participants ASAS = 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 70 = 70% improvement from baseline and an absolute change ≥ 20 units on a 0-100 scale (0=no disease activity, 100=high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: Weeks 4, 12 and 16
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Participants
  Week 4 (N = 38, 42) | 2 | 1
  Week 12 (N = 35, 37) | 8 | 7
  Week 16 (N = 28, 36) | 5 | 11

15. Secondary Outcome: Number of Participants Achieving ASAS 70 at Week 8
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) participants ASAS = 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 70 = 70% improvement from baseline and an absolute change ≥ 20 units on a 0-100 scale (0=no disease activity, 100=high disease activity)
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 36 | 42
Participants | 5 | 3
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.3291, Regression, Logistic; Odds Ratio (OR) = 2.130, 95% CI 2-sided [0.47 to 9.72]

16. Secondary Outcome: Change From Baseline in ASDAS CRP (Ankylosing Spondylitis Disease Activity Score-C Reactive Protein) Score at Week 4.
Description: The ASDAS-CRP was derived from back pain, duration of morning stiffness, patient global score and peripheral pain/swelling. The scores were categorized as follows : inactive disease(< 1.3), moderate (1.3 - < 2.1), high (2.1 - 3.5) and very high disease activity ( > 3.5). ASDAS CRP is calculated as follows:
  ASDAS CRP=0.12*Total Back Pain+0.06*Duration of Morning Stiffness+0.11*Patient Global+0.07*Peripheral Pain/Swelling+0.58*ln(CRP+1).
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 37 | 41
Units on a scale | -0.94 (0.12) | -0.16 (0.11)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; ANCOVA model on change from baseline ASDAS CRP score fitting baseline ASDAS CRP score as a covariate, plus treatment as a factor; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.11 to -0.44]

17. Secondary Outcome: Change From Baseline in ASDAS CRP Score at Week 8.
Description: as for outcome 16
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 41 | 42
Units on a scale | -1.21 (0.14) | -0.53 (0.14)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.0011, ANCOVA; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.09 to -0.28]

18. Secondary Outcome: Change From Baseline in ASDAS CRP Score at Weeks 12 and 16.
Description: as for outcome 16
Time Frame: Weeks 12 and 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 43
Units on scale
  Week 12 (N = 35, 36) | -1.4 (1.13) | -1.2 (1.07)
  Week 16 (N = 28, 33) | -1.6 (0.92) | -1.5 (1.02)

19. Secondary Outcome: Change From Baseline in ASDAS ESR (Ankylosing Spondylitis Disease Activity Score-Erythrocyte Sedimentation Rate) Score at Week 4.
Description: The ASDAS-ESR was derived from back pain, duration of morning stiffness, patient global score and peripheral pain/swelling. The scores were categorized as follows : inactive disease (< 1.3), moderate (1.3 - < 2.1), high (2.1 - 3.5) and very high disease activity ( > 3.5). ASDAS ESR is calculated as follows:
  ASDAS ESR=0.08*Total Back Pain+0.07*Duration of Morning Stiffness+0.11*Patient Global+0.09*Peripheral Pain/Swelling+0.29*√(ESR).
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 28 | 31
Units on a scale | -0.76 (0.12) | -0.19 (0.11)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; ANCOVA model on change from baseline ASDAS ESR score fitting baseline ASDAS ESR score as a covariate, plus treatment as a factor; Test type: Superiority or Other; p = 0.0011, ANCOVA; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.90 to -0.24]

20. Secondary Outcome: Change From Baseline in ASDAS ESR Score at Week 8.
Description: as for outcome 19
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 33 | 36
Units on a scale | -1.05 (0.16) | -0.38 (0.15)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.0037, ANCOVA; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.11 to -0.22]

21. Secondary Outcome: Change From Baseline in ASDAS ESR Score at Weeks 12 and 16.
Description: as for outcome 19
Time Frame: Weeks 12 and 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 37 | 37
Units on a scale
  Week 12 (N = 25, 32) | -1.0 (1.10) | -1.0 (1.01)
  Week 16 (N = 23, 26) | -1.3 (0.79) | -1.3 (1.21)

22. Secondary Outcome: Change in NSAID ASAS Score From Baseline to Week 16 (ETN Arm Only)
Description: as for outcome 1
Time Frame: Week 16
Population: The ITT population comprised all participants who received at least one dose of the randomized treatment. Participants were analyzed according to treatment randomized and any data recorded after entry into the escape arm were included in the analysis. This analysis was performed with the observed cases with no imputation.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group
Number analyzed (Participants) | 25
Scores on a scale | -65.93 (10.19)

23. Secondary Outcome: Change in NSAID ASAS Score From Week 8 to Week 16 (Placebo Only)
Description: as for outcome 1
Time Frame: Week 16
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 17
Scores on a scale | -39.22 (6.44)

24. Other Pre Specified Outcome: Change From Baseline in BAS-G (Bath Ankylosing Spondylitis-Global) Score at Week 4
Description: BAS-G was used to indicate the effect of disease has had on participant's well-being over the last 48 hours in a 0 (none) to 10 (very severe) point scale. Participants completed the BAS-G on a diary card following their Screening visit if they had a flare which required them to restart their NSAID. Participants were requested to complete the BAS-G upon symptom return (after stoppage of NSAIDs during screening phase) and weekly thereafter.
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 40 | 45
Units on a scale | -1.51 (0.33) | -0.21 (0.31)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; ANCOVA model on change from baseline BAS-G score fitting baseline BAS-G score as a covariate, plus treatment as a factor; Test type: Superiority or Other; p = 0.0050, ANCOVA; Mean Difference (Final Values) = -1.30, 95% CI 2-sided [-2.20 to -0.40]

25. Other Pre Specified Outcome: Change From Baseline in BAS-G Score at Week 8
Description: as for outcome 24
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 41 | 45
Units on a scale | -2.29 (0.40) | -1.05 (0.38)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.0256, ANCOVA; Mean Difference (Final Values) = -1.24, 95% CI 2-sided [-2.33 to -0.16]

26. Other Pre Specified Outcome: Change From Baseline in BAS-G Score at Weeks 12 and 16.
Description: as for outcome 24
Time Frame: Weeks 12 and 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Units on a scale
  Week 12 (N = 36, 41) | -2.8 (2.50) | -2.4 (2.72)
  Week 16 (N = 28, 36) | -2.6 (2.08) | -2.6 (3.12)

27. Other Pre Specified Outcome: Change From Baseline in Total Back Pain at Week 4
Description: Participants assessed the total back pain they had in the previous 48 hours on a scale from 0 (no pain) to 10 (most severe pain).
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 40 | 45
Units on a scale | -1.59 (0.36) | -0.58 (0.34)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; ANCOVA model on change from baseline total back pain fitting baseline total back pain as a covariate, plus treatment as a factor; Test type: Superiority or Other; p = 0.0474, ANCOVA; Mean Difference (Final Values) = -1.01, 95% CI 2-sided [-2.00 to -0.01]

28. Other Pre Specified Outcome: Change From Baseline in Total Back Pain at Week 8
Description: as for outcome 27
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 41 | 45
Units on a scale | -2.24 (0.39) | -0.96 (0.37)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p = 0.0212, ANCOVA; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-2.36 to -0.20]

29. Other Pre Specified Outcome: Change From Baseline in Total Back Pain at Weeks 4, 8, 12 and 16
Description: as for outcome 27
Time Frame: Weeks 4, 8, 12 and 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Units on a scale
  Week 4 (N = 40, 45) | -1.1 (2.10) | -0.3 (1.32)
  Week 8 (N = 37, 43) | -1.7 (2.28) | -0.8 (1.72)
  Week 12 (N= 36, 42) | -2.6 (2.62) | -2.6 (2.34)
  Week 16 (N = 28, 37) | -2.9 (2.17) | -2.6 (2.33)

30. Other Pre Specified Outcome: Change From Baseline in Nocturnal Back Pain at Week 4
Description: Participants assessed the nocturnal back pain they had in the previous 48 hours on a scale from 0 (no pain) to 10 (most severe pain).
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 40 | 45
Units on a scale | -2.13 (0.40) | -0.82 (0.38)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; ANCOVA model on change from baseline nocturnal back pain fitting baseline nocturnal back pain as a covariate, plus treatment as a factor; Test type: Superiority or Other; p = 0.0198, ANCOVA; Mean Difference (Final Values) = -1.31, 95% CI 2-sided [-2.40 to -0.21]

31. Other Pre Specified Outcome: Change From Baseline in Nocturnal Back Pain at Week 8
Description: as for outcome 30
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 41 | 45
Units on a scale | -2.71 (0.43) | -1.20 (0.41)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; [analysis description as in outcome 30, analysis 1]; Test type: Superiority or Other; p = 0.0132, ANCOVA; Mean Difference (Final Values) = -1.51, 95% CI 2-sided [-2.69 to -0.32]

32. Other Pre Specified Outcome: Change From Baseline in Nocturnal Back Pain at Weeks 12 and 16
Description: as for outcome 30
Time Frame: Weeks 12 and 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Units on a scale
  Week 12 (N = 36, 42) | -3.0 (2.88) | -3.0 (2.98)
  Week 16 (N = 28, 37) | -2.9 (2.14) | -3.5 (2.72)

33. Other Pre Specified Outcome: Change From Baseline in BASFI (Bath Ankylosing Spondylitis Functional Index ) at Week 4
Description: Participants assessed their level of ability to complete activities on a scale from 0 (easy) to 10 (impossible). These scales were collected at each visit in the CRF. The total score was calculated as the average score of the 10 questions.
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 40 | 45
Units on a scale | -1.13 (0.25) | -0.32 (0.24)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; ANCOVA model on change from baseline BASFI score fitting baseline BASFI score as a covariate, plus treatment as a factor; Test type: Superiority or Other; p = 0.0237, ANCOVA; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.50 to -0.11]

34. Other Pre Specified Outcome: Change From Baseline in BASFI at Week 8
Description: as for outcome 33
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 41 | 45
Units on a scale | -1.68 (0.30) | -0.77 (0.29)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; [analysis description as in outcome 33, analysis 1]; Test type: Superiority or Other; p = 0.0297, ANCOVA; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-1.74 to -0.09]

35. Other Pre Specified Outcome: Change From Baseline in BASDAI Level of Morning Stiffness-related Scores at Week 4
Description: Participants were requested to complete the BASDAI upon symptom return then every day for the first 15 days after first administration of test article and weekly thereafter. A numeric rating scale was used, for questions 1-5 (Fatigue, Spinal Pain, Joint pain or swelling, discomfort and morning stiffness severity respectively) it was on the scale from 0 (none) to 10 (very severe). For question 6 (morning stiffness duration) it was on the scale of 0 (0 or more hours) to 10 (2 hours). The analysis presented below is the change in morning stiffness severity.
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 39 | 44
Units on a scale | -2.23 (0.34) | -1.07 (0.32)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; ANCOVA model on change from each baseline BASDAI component score fitting each baseline component score as a covariate, plus treatment as a factor; Test type: Superiority or Other; p = 0.0152, ANCOVA; Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-2.09 to -0.23]

36. Secondary Outcome: Change From Baseline in BASDAI Level of Morning Stiffness-related Scores at Week 8
Description: as for outcome 35
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 41 | 45
Units on a scale | -2.74 (0.39) | -1.59 (0.37)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; [analysis description as in outcome 35, analysis 1]; Test type: Superiority or Other; p = 0.0344, ANCOVA; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-2.22 to -0.09]

37. Other Pre Specified Outcome: Change From Baseline in BASDAI Level of Morning Stiffness-related Scores at Weeks 12 and 16
Description: as for outcome 35
Time Frame: Weeks 12 and 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Units on a scale
  Week 12 (N = 36, 42) | -3.4 (2.75) | -3.0 (2.74)
  Weel 16 (N = 28, 37) | -3.3 (2.64) | -3.9 (2.46)

38. Other Pre Specified Outcome: Change From Baseline in PGA (Physician Global Assessment) at Week 4
Description: The investigator assessed the overall disease activity using the scale of 0 (no disease activity) to 10 (severe disease activity).
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 40 | 44
Units on a scale | -2.05 (0.30) | -0.71 (0.28)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; ANCOVA model on change from baseline PGA score fitting baseline PGA score as a covariate, plus treatment as a factor; Test type: Superiority or Other; p = 0.0017, ANCOVA; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-2.16 to -0.52]

39. Other Pre Specified Outcome: Change From Baseline in PGA (Physician Global Assessment) at Week 8
Description: Investigator assessed the overall disease activity using the scale of 0 (no disease activity) to 10 (severe disease activity).
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 40 | 44
Units on a scale | -2.69 (0.35) | -1.58 (0.33)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; ANCOVA model on change from baseline PGA score fitting baseline PGA score as a covariate, plus treatment as a factor; Test type: Superiority or Other; p = 0.0233, ANCOVA; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-2.07 to -0.16]

40. Other Pre Specified Outcome: Change From Baseline in PGA at Weeks 12 and 16
Description: as for outcome 39
Time Frame: Weeks 12 and 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 41 | 46
Units on a scale
  Week 12 (N = 35, 38) | -3.5 (2.73) | -3.4 (1.54)
  Week 16 (N = 29, 37) | -3.7 (2.22) | -3.8 (2.00)

41. Other Pre Specified Outcome: Change From Baseline in Each BASFI Component at Week 4
Description: BASFI is to assess the prticipant's level of ability to complete the activities on a scale from 0 (easy) to 10 (impossible). The total score was calculated as the average score of the 10 questions.
Time Frame: Week 4
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Units on a scale
  Putting on socks (N = 40, 45) | -1.0 (2.66) | -0.4 (1.72)
  Bending forward (N = 40, 45) | -1.0 (3.19) | -0.2 (1.96)
  Reaching up high (N = 40, 45) | -1.3 (2.43) | -0.3 (1.62)
  Getting out of an armless chair (N = 40, 45) | -1.3 (2.58) | -0.5 (1.69)
  Getting up off floor from back (N = 40, 45) | -1.6 (2.91) | -0.4 (1.69)
  Standing unsupported 10 min (N = 40, 45) | -1.0 (2.57) | 0.0 (2.57)
  Climbing steps without aid (N = 40, 45) | -0.4 (3.00) | -0.5 (2.04)
  Looking over shoulder | -1.6 (2.70) | -0.2 (2.15)
  Physically demanding activities (N = 40, 45) | -1.2 (2.34) | -0.4 (1.93)
  Full day's activities (N = 40, 45) | -1.1 (2.42) | -0.4 (1.75)

42. Other Pre Specified Outcome: Change From Baseline in Each BASFI Component at Week 8
Description: as for outcome 41
Time Frame: Week 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Units on a scale
  Putting on socks (N = 37, 43) | -1.3 (2.64) | -0.3 (2.18)
  Bending forward (N = 37, 43) | -1.8 (3.10) | -0.4 (2.08)
  Reaching up high (N = 37, 43) | -1.3 (3.09) | -0.7 (2.02)
  Getting out of an armless chair (N = 37, 43) | -2.1 (2.78) | -1.0 (2.23)
  Getting up off floor from back (N = 37, 43) | -2.3 (3.01) | -0.6 (2.33)
  Standing unsupported 10 min (N = 37, 43) | -1.6 (2.66) | -0.8 (2.67)
  Climbing steps without aid (N = 37, 43) | -1.2 (3.22) | -0.9 (2.26)
  Looking over shoulder (N = 37, 43) | -2.4 (2.79) | -0.8 (1.71)
  Physically demanding activities (N = 37, 41) | -1.8 (2.11) | -1.2 (1.91)
  Full day's activities (N = 37, 41) | -1.4 (2.63) | -1.2 (2.04)

43. Other Pre Specified Outcome: Change From Baseline in Each BASFI Component at Week 12
Description: as for outcome 41
Time Frame: Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Units on a scale
  Putting on socks (n = 36, 42) | -1.6 (2.75) | -1.6 (2.39)
  Bending forward (N = 36, 42) | -2.2 (3.25) | -1.7 (2.56)
  Reaching up high (N = 36,42) | -1.7 (3.21) | -1.5 (2.35)
  Getting out of an armless chair (N = 36, 42) | -2.6 (3.38) | -2.0 (2.50)
  Getting up off floor from back (N = 36, 42) | -2.5 (3.09) | -1.7 (2.66)
  standing unsupported 10 min (N = 36,42) | -2.0 (2.49) | -2.1 (2.95)
  Climbing steps without aid (N = 36, 42) | -1.6 (3.18) | -1.4 (2.43)
  Looking over shoulder (N = 36, 42) | -2.6 (2.92) | -1.8 (2.62)
  Physically demanding activities (N = 36, 41) | -2.2 (2.68) | -2.3 (2.29)
  Full day's activities (N = 36, 40) | -1.8 (2.45) | -2.3 (2.12)

44. Other Pre Specified Outcome: Change From Baseline in Each BASFI Component at Week 16
Description: as for outcome 41
Time Frame: Week 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Units on a scale
  Putting on socks (N = 28, 37) | -1.1 (3.18) | -2.1 (2.40)
  Bending forward (N = 28, 37) | -2.0 (3.36) | -2.1 (2.33)
  Reaching up high (N = 27, 37) | -1.0 (3.55) | -1.6 (2.29)
  Getting out of an armless chair (N = 28, 37) | -2.0 (3.42) | -2.5 (2.35)
  Getting up off floor from back (N = 28, 37) | -2.2 (2.83) | -2.3 (2.60)
  Standing unsupported 10 min (N = 28, 37) | -2.2 (2.5) | -2.6 (2.8)
  Climbing steps without aid (N = 28, 37) | -1.3 (3.13) | -1.9 (2.53)
  Looking over shoulder (N = 28, 37) | -2.4 (3.19) | -2.3 (2.62)
  Physically demanding activities (N = 28, 36) | -2.3 (2.46) | -2.6 (2.38)
  Full day's activities (N = 28, 36) | -1.9 (2.28) | -2.6 (2.07)

45. Other Pre Specified Outcome: Change From Baseline in Swollen Joint Counts at Weeks 4, 8, 12 and 16
Description: Swollen joint count was performed at each visit to assess the peripheral joint involvement according to ASAS recommendation.
Time Frame: Weeks 4, 8, 12 and 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Swollen joints
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 28 | 35
Swollen joints
  Week 4 (N = 23, 22) | -0.6 (1.65) | 0.0 (1.09)
  Week 8 (N = 14, 22) | -0.1 (2.09) | 0.0 (1.25)
  Weel 12 (N = 11, 15) | -0.5 (1.29) | -0.3 (1.23)
  Week 16 (N = 9, 9) | -1.1 (2.89) | 2.3 (6.65)

46. Other Pre Specified Outcome: Change From Baseline in Tenderness Joint Counts at Weeks 4, 8, 12 and 16
Description: Tender joint count was performed at each visit to assess the peripheral joint involvement according to ASAS recommendation.
Time Frame: Weeks 4, 8, 12 and 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Tender joints
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 28 | 35
Tender joints
  Week 4 (N = 23, 22) | -1.2 (3.61) | -2.4 (7.57)
  Week 8 (N = 14, 22) | -2.3 (5.11) | -3.1 (6.47)
  Week 12 (N = 11, 15) | -1.3 (5.00) | -1.4 (10.70)
  Week 16 (N = 9, 9) | -1.9 (5.64) | 0.2 (9.93)

47. Other Pre Specified Outcome: Change From Baseline in MASES (Maastricht Ankylosing Spondylitis Entheses Score) Score at Weeks 4, 8, 12 and 16
Description: Assessment of enthesitis was performed in the following 7 domains: 1) 1st costochondral joint left and right, 2) 7th costochondral joint left and right, 3) posterior superior iliac spine left and right, 4) anterior superior iliac spine left and right, 5) iliac crest left and right, 6) 5th lumbar spinous process and 7) proximal insertion of Achilles tendon left and right. Each domain was graded for the presence (1) and absence (0) of tenderness yielding total MASES ranging from 0 (no tenderness) to 13 (worst possible score; severe tenderness).
Time Frame: Weeks 4, 8, 12 and 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 35 | 35
Units on a scale
  Week 4 (N = 23, 27) | -0.7 (2.55) | -0.3 (2.31)
  Week 8 (N = 20, 24) | -1.1 (2.42) | -0.7 (2.55)
  Week 12 (N = 14, 13) | -1.0 (2.94) | 0.0 (2.77)
  Week 16 (N = 13, 10) | -0.6 (2.57) | -1.4 (3.27)

48. Other Pre Specified Outcome: Number of Participants With Minimum Clinically Important Improvement (MCII) at Week 8
Description: MCII was completed at visit weeks 4, 8, 12 and 16 or Early Discontinuation and once weekly between visits. MCII was converted to binary scores as follows: 1 = 'improved'/'very important' and 'improved'/'moderately important' 2 = 'improved'/'slightly important', 'improved'/'not at all important', 'no change' and 'worse-no pain'. MCII was determined based on participant's response on the following three items for the question of how have they been during the last 48 hours compared to when they started the study: improved or less pain, no change and worse-more pain. MCII was typically defined according to the patients perception of what was very important improvement, moderate important improvement, slightly important improvement or not at all improvement.
Time Frame: Week 8
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 37 | 43
Participants | 21 | 17
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; Week 8 was analyzed using logistic regression with baseline score and treatment group included as covariates; Test type: Superiority or Other; p = 0.1260, Regression, Logistic; Odds Ratio (OR) = 2.01, 95% CI 2-sided [0.822 to 4.901]

49. Other Pre Specified Outcome: Number of Participants With MCII at Weeks 4, 12 and 16
Description: MCII was completed at Weeks 4, 8, 12 and 16 or Early Discontinuation and once weekly between visits. MCII was converted to binary scores as follows: 1 = 'improved'/'very important' and 'improved'/'moderately important' 2 = 'improved'/'slightly important', 'improved'/'not at all important', 'no change' and 'worse-no pain. MCII was determined based on participant's response on the following three items for the question of how have they been during the last 48 hours compared to when they started the study: improved or less pain, no change and worse-more pain. MCII was typically defined according to the patients perception of what was very important improvement, moderate important improvement, slightly important improvement or not at all improvement.
Time Frame: Weeks 4, 12 and 16
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Participants
  Week 4 (N = 40, 44) | 19 | 11
  Week 12 (N = 36, 42) | 25 | 25
  Week 16 (N = 28, 37) | 22 | 22

50. Other Pre Specified Outcome: Number of Participants With Minimum Clinically Important Deterioration (MCID) at Weeks 4, 8, 12 and 16
Description: MCID was completed at Weeks 4, 8, 12 and 16 or Early Discontinuation and once weekly between visits. MCID was converted to binary scores as follows: 1 = 'improved'/'very important' and 'improved'/'moderately important' 2 = 'improved'/'slightly important', 'improved'/'not at all important', 'no change' and 'worse-no pain. MCID was evaluated based on participant's opinion on the following three items for the question of how have they been during the last 48 hours compared to Screening visit: 'improved-less pain', 'no change', and 'worse-more pain'. Participants were further asked the importance of worsening i.e., very important, moderately important, slightly important and not at all important as MCID evaluation criteria.
Time Frame: Weeks 4, 8, 12 and 16
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Participants
  Week 4 (N = 40, 44) | 3 | 9
  Week 8 (N = 37, 43) | 0 | 3
  Week 12 (N = 36, 42) | 0 | 0
  Week 16 (N = 28, 37) | 0 | 0

51. Other Pre Specified Outcome: Number of Participants With Patient Acceptable Symptom State (PASS) at Week 8
Description: PASS is defined as a symptom state that the participants consider acceptable. PASS was collected weekly in the diary card, but at each visit this was collected in the CRF. Participants assessed their health in the previous 48 hours and whether it would be acceptable to remain like that in the next few months.
Time Frame: Week 8
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 37 | 43
Participants | 22 | 16
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; Logistic regression with baseline morning stiffness score and treatment group included as covariates. Week 8 was analyzed using a logistic regression to assess treatment effect; Test type: Superiority or Other; p = 0.0498, Regression, Logistic; Odds Ratio (OR) = 2.47, 95% CI 2-sided [1.00 to 6.08]

52. Other Pre Specified Outcome: Number of Participants With PASS at Weeks 4, 12 and 16
Description: PASS is defined as a symptom state that the participants consider acceptable. The PASS was collected weekly in the diary card, but at each visit this was collected in the CRF. Participants assessed their health in the previous 48 hours and whether it would be acceptable to remain like that in the next few months.
Time Frame: Weeks 4, 12 and 16
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Participants
  Week 4 (N = 40, 44) | 19 | 14
  Week 12 (N = 36, 42) | 23 | 29
  Week 16 (N = 28, 37) | 20 | 28

53. Other Pre Specified Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) at Week 4
Description: BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: cervical rotation, intermalleolar distance, modified Schober's test, lateral flexion and tragus to wall distance. Each measure was scored 0-2 (0=normal mobility, 2=severe reduction) to give a final score ranging 0 to 10.
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 39 | 45
Units on a scale | -0.31 (0.19) | 0.05 (0.17)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; ANCOVA model on change from baseline BASMI score fitting baseline BASMI score as a covariate, plus treatment as a factor; Test type: Superiority or Other; p = 0.1601, ANCOVA; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.87 to 0.15]

54. Other Pre Specified Outcome: Change From Baseline in BASMI at Week 8
Description: as for outcome 53
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 40 | 46
Units on a scale | -0.40 (0.21) | -0.11 (0.19)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; [analysis description as in outcome 53, analysis 1]; Test type: Superiority or Other; p = 0.2967, ANCOVA; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.86 to 0.27]

55. Other Pre Specified Outcome: Change From Baseline in BASMI at Weeks 12 and 16
Description: as for outcome 53
Time Frame: Weeks 12 and 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 41 | 48
Units on a scale
  Week 12 (N = 35, 43) | -0.4 (1.44) | -0.4 (1.26)
  Week 16 (N = 28, 38) | -0.6 (1.71) | -0.6 (1.23)

56. Other Pre Specified Outcome: Change From Baseline in BASMI Components at Week 4
Description: BASMI is an objective measure of spinal mobility. The BASMI score was composed of 5 measures: cervical rotation, intermalleolar distance, modified Schober's test, lateral flexion and tragus to wall distance. Each measure was scored 0-2 (0=normal mobility, 2=severe reduction) to give a final score ranging 0 to 10. For each BASMI component, the best of the two tries was taken which corresponded to the highest value for cervical rotation, intermalleolar distance, modified Schober's test and lateral flexion and the smallest value for tragus to wall distance. For cervical rotation, lateral flexion and tragus to wall distance, a mean of the left and right measurements was taken.
Time Frame: Week 4
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Units on a scale
  Cervical rotation (N = 39, 45) | 0.0 (0.46) | 0.0 (0.34)
  Tragus to wall distance (N=41, 43) | 0.0 (0.31) | 0.0 (0.49)
  Lateral flexion (N = 40, 42) | -0.1 (0.61) | -0.1 (0.50)
  Modified schober's test (N = 41, 45) | 0.0 (0.55) | 0.1 (0.68)
  Intermalleolar distance (N = 38, 44) | -0.2 (0.73) | 0.1 (0.66)

57. Other Pre Specified Outcome: Change From Baseline in BASMI Components at Week 8
Description: as for outcome 56
Time Frame: Week 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Units on a scale
  Cervical rotation (N = 37, 44) | -0.1 (0.60) | 0.0 (0.53)
  Tragus to wall distance (N = 38, 43) | 0.1 (0.40) | -0.1 (0.43)
  Lateral flexion (N = 38, 42) | -0.1 (0.58) | -0.1 (0.55)
  Modified schober's test (N = 38, 44) | -0.1 (0.54) | 0.1 (0.67)
  Intermalleolar distance (N = 36, 43) | -0.2 (0.75) | 0.0 (0.76)

58. Other Pre Specified Outcome: Change From Baseline in BASMI Components at Week 12
Description: as for outcome 56
Time Frame: Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Units on a scale
  Cervical rotation (N= 35, 43) | -0.1 (0.66) | -0.1 (0.40)
  Tragus to wall distance (N = 36, 42) | 0.2 (0.51) | 0.0 (0.41)
  Lateral flexion (N = 36, 42) | -0.2 (0.56) | -0.2 (0.40)
  Modified schober's test (N = 36, 43) | -0.1 (0.55) | 0.0 (0.77)
  Intermalleolar distance (N = 33, 42) | -0.2 (0.88) | -0.1 (0.77)

59. Other Pre Specified Outcome: Change From Baseline in BASMI Components at Week 16
Description: as for outcome 56
Time Frame: Week 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 42 | 48
Units on a scale
  Cervical rotation (N = 28, 38) | -0.1 (0.54) | -0.1 (0.56)
  Tragus to wall distance (N = 29, 37) | 0.0 (0.33) | -0.1 (0.47)
  Lateral flexion (N= 29, 36) | -0.1 (0.64) | -0.2 (0.47)
  Modified schober's test (N = 29, 38) | -0.1 (0.49) | 0.0 (0.77)
  Intermalleolar distance (N = 26, 37) | -0.3 (0.87) | -0.2 (0.66)

60. Other Pre Specified Outcome: Change From Baseline in Chest Expansion at Week 4
Description: Chest expansion, measured in cm, is defined as the difference in thoracic circumference during full expiration versus full inspiration, measured at the fourth intercostal space (nipple line). Chest expansion was measured for both maximum and minimum inhalation and the data presented below combined both the values.
Time Frame: Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 37 | 44
cm | 2.61 (1.61) | 0.21 (1.48)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; ANCOVA model on change from baseline in chest expansion mobility score fitting baseline chest expansion mobility score as a covariate, plus treatment as a factor; Test type: Superiority or Other; p = 0.2735, ANCOVA; Mean Difference (Final Values) = 2.41, 95% CI 2-sided [-1.94 to 6.75]

61. Other Pre Specified Outcome: Change From Baseline in Chest Expansion at Week 8
Description: as for outcome 60
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 39 | 45
cm | 0.62 (0.24) | -0.06 (0.23)
Statistical Analysis 1: Comparison: Double Blind ETN 50 mg to Open Label ETN 50 mg Group vs Placebo to Open Label ETN 50 mg Group; [analysis description as in outcome 60, analysis 1]; Test type: Superiority or Other; p = 0.0422, ANCOVA; Mean Difference (Final Values) = 0.68, 95% CI 2-sided [0.02 to 1.34]

62. Other Pre Specified Outcome: Change From Baseline in Chest Expansion at Weeks 12 and 16
Description: as for outcome 60
Time Frame: Weeks 12 and 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Number analyzed (Participants) | 40 | 47
cm
  Week 12 (N = 34, 42) | 0.3 (2.26) | 0.1 (2.03)
  Week 16 (N = 27, 37) | 0.2 (1.42) | 2.0 (10.92)

ADVERSE EVENTS:
Time Frame: Up to Week 16 and safety follow-up at 4 weeks after the last visit
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Double Blind ETN 50 mg to Open Label ETN 50 mg Group | Placebo to Open Label ETN 50 mg Group
Serious Adverse Events (participants affected / at risk) | 1/42 | 2/48
Other Adverse Events (participants affected / at risk) | 34/42 | 34/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind ETN 50 mg to Open Label ETN 50 mg Group (N=42) | Placebo to Open Label ETN 50 mg Group (N=48)
Duodenitis (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Cyst Removal (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind ETN 50 mg to Open Label ETN 50 mg Group (N=42) | Placebo to Open Label ETN 50 mg Group (N=48)
Palpitations (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Dry Eye (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Gastric Disorder (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 3 | 4
Condition Aggravated (General disorders) | 1 | 0
Injection Site Erythema (General disorders) | 2 | 4
Injection Site Hypersensitivity (General disorders) | 3 | 0
Injection Site Pain (General disorders) | 1 | 0
Injection Site Pruritus (General disorders) | 2 | 2
Injection Site Reaction (General disorders) | 3 | 3
Fatigue (General disorders) | 0 | 1
Infusion Site Erythema (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1
Hepatocellular Injury (Hepatobiliary disorders) | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Ear Infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gingivitis (Infections and infestations) | 1 | 0
Nail Infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 4
Oral Herpes (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 1 | 2
Rhinitis (Infections and infestations) | 5 | 3
Sinusitis (Infections and infestations) | 1 | 0
Tooth Infection (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 2 | 0
Viral Infection (Infections and infestations) | 1 | 0
Viral Rhinitis (Infections and infestations) | 1 | 1
Escherichia Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 3
Pyelonephritis (Infections and infestations) | 0 | 1
Tooth Abscess (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 2
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 1
Inappropriate Schedule Of Drug Administration (Injury, poisoning and procedural complications) | 1 | 0
Incision Site Pain (Injury, poisoning and procedural complications) | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0
Medication Error (Injury, poisoning and procedural complications) | 1 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 2
Blood Glucose Increased (Investigations) | 1 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Blood Cholesterol Increased (Investigations) | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 1
Glycosylated Haemoglobin Increased (Investigations) | 0 | 1
Platelet Count Decreased (Investigations) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 5 | 3
Migraine (Nervous system disorders) | 2 | 0
Presyncope (Nervous system disorders) | 1 | 0
Aphonia (Nervous system disorders) | 0 | 1
Initial Insomnia (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Sleep Disorder (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis Seasonal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Allergic Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Skin Plaque (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Tooth Extraction (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 1 | 2
Flushing (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.